CLINICAL TRIAL: NCT04361513
Title: Genicular Nerve Block in Rheumatoid Arthritis: a Prospective Randomized Clinical Trial
Brief Title: Genicular Nerve Block in Rheuamtoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Associate professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28/4/2020
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Pain; Joint Function Disorder; Inflammation
MeSH Terms: conditions — Pain; Inflammation | interventions — Bupivacaine; Triamcinolone

STUDY DESIGN:
Intervention Model Description: Group received nerve block and another group received steroid
Who Masked: Participant
Masking Description: The participants does not know the nature of the injected material. Syringe was colored to cover it
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve block group (Active Comparator): 3 point genicular nerve block under ultrasound guidance. half ml of Bupivacaine hydrochloride 0.5% (Marcaine, Pfizer) was injected in each point.
  Interventions: Drug: Bupivacaine hydrochloride 0.5% (Marcaine, Pfizer); Drug: triamcinolone 40 milligrams (Kenacort, Bristol Myers Squip)
- intra-articular steroid injection (Other): 1 mL of triamcinolone 40 milligrams (Kenacort, Bristol Myers Squip) was injected intraarticular.
  Interventions: Drug: Bupivacaine hydrochloride 0.5% (Marcaine, Pfizer); Drug: triamcinolone 40 milligrams (Kenacort, Bristol Myers Squip)

INTERVENTIONS:
Drug: Bupivacaine hydrochloride 0.5% (Marcaine, Pfizer) — 3 point genicular nerve block
Drug: triamcinolone 40 milligrams (Kenacort, Bristol Myers Squip) — intra-articular injection of triamcinilone

SUMMARY:
N=64 RA patients either early or established disease diagnosed after ACR/EULAR criteria 2010 with unilateral persistent knee arthritis. They were randomly assigned into two groups; group 1 received genicular nerve block, group 2 intra-articular triamcinolone. Both groups were examined by SOLAR scoring system, Visual analogue scale (VAS) and Lysholm score at 0, 2 and 12 weeks. A semi-quantitative score was used to assess tenderness and swelling at the same intervals.

ELIGIBILITY:
Inclusion Criteria:

* RA patients
* Age > 18
* unilateral persistent knee arthritis

Exclusion Criteria:

* Participants with severe knee osteoarthritis
* peripheral neuropathy
* psoriatic arthritis
* skin infection
* or those who have allergy for Bupivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Pain changes by VAS | at 0 time after 2 weeks and after 12 weeks
  0 means no pain and 10 means the most severe pain
SOLAR score for inflammation changes by ultrasound | at 0 time after 2 weeks and after 12 weeks
  0 means normal and 27 means the worst possible inflammation
Lysholm score for change in knee function | at 0 time after 2 weeks and after 12 weeks
  100 means the best performance and 0 means complete loss of function

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university, Minya, Egypt